CLINICAL TRIAL: NCT05290220
Title: An Open-label, Multicenter, Phase II Clinical Study to Evaluate the Efficacy and Safety of HLX07 (A Recombinant Humanized Anti-EGFR Monoclonal Antibody Injection) Combination Therapy or Motherapy in Patient With Advanced Hepatocellular Carcinoma (HCC)
Brief Title: HLX07 Combination Therapy or Motherapy in Patient With Advanced Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HLX07-HCC201
Record Dates: First submitted 2022-03-07; First posted 2022-03-22 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-03

CONDITIONS: Advanced Hepatocellular Carcinoma
MeSH Terms: interventions — HLX07; lenvatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A: As first-line therapy (Experimental): HLX07 1500 mg + HLX10 300 mg + HLX04 15mg/kg iv q3w
  Interventions: Drug: HLX07; Drug: HLX10; Drug: HLX04
- Arm B: As second-line therapy (Experimental): HLX07 1500 mg iv Q3w + Lenvatinib 12 mg (BW≥60 kg) or 8 mg (BW <60 kg) po qd
  Interventions: Drug: HLX07; Drug: lenvatinib
- Arm C:As third-line or above therapy (Experimental): HLX07 1500 mg iv Q3w
  Interventions: Drug: HLX07

INTERVENTIONS:
Drug: HLX07 — 1500 mg
Drug: HLX10 — 300 mg
  Arms: Arm A: As first-line therapy
Drug: HLX04 — 15mg/kg
  Arms: Arm A: As first-line therapy
Drug: lenvatinib — 12 mg (BW≥60 kg) or 8 mg (BW <60 kg)
  Arms: Arm B: As second-line therapy

SUMMARY:
This study is conducted in patients with advanced hepatocellular carcinoma (HCC). This study includes three arms: A, B, and C. Arm A will receive HLX07 combination therapy with HLX10 and HLX04 as first line treatment. Arm B will receive HLX07 combination therapy with lenvatinib as second line treatment. Arm C will receive HLX07 monotherapy as third-line or above treatment. All of eligible patients will receive study drug treatment until loss of clinical benefit, unacceptable toxicity, death, withdrawal of informed consent (whichever occurs first, HLX10 treatment up to 2 years).

ELIGIBILITY:
Inclusion Criteria:

Subjects who meet all of the following criteria are allowed to be enrolled into this study:

1. Volunteer to participate in this clinical study; completely understand and know this study as well as sign the informed consent form (ICF); be willing to follow and be able to complete all study procedures.
2. Age ≥ 18 years and ≤ 75 years when ICF is signed.
3. Histopathologically or cytologically confirmed diagnosis of advanced hepatocellular carcinoma (HCC), Or the clinical diagnosis meets the american association for the study of liver diseases (AASLD) diagnostic criteria for HCC.
4. prior therapy: Arm A: Never received systemic anti-tumor drug therapy before. Arm B: Patient has a contraindication or intolerance to, or has failed treatment with 1-line systemic anti-tumor therapy (PD-1 /L1 -based combination therapies). Arm C: Previously received second or greater lines of systemic therapy. （Including： 1. PD-1/L1-based therapy 2. Lenvatinib or Sorafenib).
5. According to the curative effect evaluation criteria in solid tumors (RECIST) v1.1, assessed by the investigator with at least one measurable lesions. Measurable target lesions cannot be selected from the site of previous radiotherapy.

   (lesions located in the usual radiation area, if confirm progress, can also be selected as the target lesion).
6. Child-pugh liver function rating within 7 days before the first administration of the study drug : grade A and good grade B (≤ 7 points).
7. Arm B,C: The end of previous systematic treatment() must be ≥ 2 weeks before the first administration of the study drug, and the treatment-related AE should be restored to the level of NCI -CTCAE ≤ 1 (except hair loss).
8. The patient with HCC has liver surgery or local treatment (hepatic artery embolization, TACE, hepatic artery infusion, radiofrequency ablation, cryoablation or percutaneous ethanol injection) , Arm A and B : treatment was received ≥ 4 weeks prior to the first administration of this study. Arm C: treatment was received ≥ 2 weeks prior to the first administration of this study; The palliative radiotherapy for bone metastases was received ≥ 2 weeks prior to the first administration of this study; The diagnostic liver puncturewas received ≥ 1weeks prior to the first administration of this study. AEs related to previous local therapy should be recovered to the level of NCI -CTCAE ≤ 1.
9. The ECOG physical performance score within 7 days before the first administration of the study drug was 0 or 1.
10. Expected survival ≥ 12 weeks.
11. If HBsAg (+) or HBcAb (+), HBV-DNA must be<2500 copy/ml or ≤ 500 IU/mL or <ULN to be included in the group, and those with elevated HBV-DNA must agree to receive nucleoside anti-hepatitis b virus treatment. Subjects with negative HCV antibody (-) or HCV-RNA were admitted. If HCV-RNA is positive, must agree to receive standard of anti-virus treatment, and subjects must have ALT and AST ≤ 3×ULN to be enrolled. Subjects with co-infection of hepatitis b and c should be excluded.
12. The functions of the vital organs meet the following requirements (no blood transfusion, albumin, colony-stimulating factor, or platelet raising drugs are allowed within 14 days before the first use of the study drugs); Absolute neutrophil count (ANC) ≥1.5×109/L platelet≥ 100×109/L; Hemoglobin≥ 90g/ L; Serum albumin≥ 30g/L; Total bilirubin≤ 1.5 ULN, ALT, AST≤ 5 ULN(exclude the HCV-RNA is positive patients);Serum creatinine≤1.5 ULN or creatinine clearance > 50 mL/min (Cockcroft-Gault formula);APTT, INR and PT ≤1.5 ULN; Qualitative analysis of proteinuria≤1+; If ≥2+, 24-hour urine protein test is required, and the subject must have<1g to be enrolled.
13. For fertile female subjects, the serum pregnancy test must be negative within 7 days before the first dose.Subject agrees to use effective contraception.

Exclusion Criteria:

Subjects who meet any of the following criteria are not allowed to be enrolled in this study:

1. Hepatobiliary duct cell carcinoma, mixed cell carcinoma, or fibroblastic layer cell carcinoma are known.
2. Hepatic encephalopathy within 6 months before the first administration of the study drug.
3. According to the images, portal vein invasion, inferior vena cava or cardiac involvement of HCC main portal branch (Vp4) were present. Patients with cancer thrombus in main portal vein but smooth blood flow in contralateral branch can be enrolled.
4. Other active malignancies within 3 years prior to the first administration of the study drug.Curable localized tumors, such as basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder carcinoma, carcinoma in situ of the prostate, cervical carcinoma in situ, and carcinoma in situ of the breast, can be included in the group.
5. People who are ready to undergo or have received organ or bone marrow transplants.
6. After appropriate intervention, uncontrollable pleural effusion, pericardial effusion or ascites still need to be drained frequently (once a month or more frequently).
7. Symptomatic brain or meningeal metastases (unless the patient has been on > treatment for 3 months, has no evidence of progress on imaging within 4 weeks prior to initial administration, and tumor-related clinical symptoms are stable).
8. Cerebrovascular accident, Pulmonary embolism, deep vein thrombosis or any other serious thromboembolism, myocardial infarction, unstable angina pectoris and poorly controlled arrhythmia occurred within half a year (including QTc interval ≥ 450 ms for men and ≥ 470 ms for women) (QTc interval was calculated by Fridericia formula).
9. According to the New York heart association (NYHA) standard levels Ⅲ or Ⅳ cardiac insufficiency or heart colour to exceed examination: LVEF(left ventricular ejection fraction) < 50%.
10. Human immunodeficiency virus (HIV) infection.
11. Active tuberculosis.Patients with previous and current cases of interstitial pneumonia, pneumoconiosis, radioactive pneumonia, drug-related pneumonia, and severe impairment of lung function that may interfere with the detection and management of suspected drug-related lung toxicity.
12. Within 14 days prior to the first administration of the study drug, any active infection requiring systematic anti-infective treatment occurs.
13. Major surgery was performed within 28 days prior to the first administration of the study drug. Major surgery in this study was defined as the minimum recovery time of 3 weeks after surgery before the surgery treated in this study could be performed.
14. Within 14 days prior to the first administration of the study drug, participating in other clinical studies.
15. Subjects requiring systemic treatment with corticosteroids (> 10 mg/ day or equivalent dose of prednisone) or other immunosuppressants within 14 days prior to or during the study.In the absence of active autoimmune disease, the inhalation or topical use of steroids, or adrenal hormone replacement at doses less than 10 mg/ day of prednisone efficacy, is permitted.
16. Patients who have previously received systemic anti-EGFR monoclonal antibody therapy.
17. History of severe hypersensitivity to any monoclonal antibody or study drug excipient.
18. Pregnant or lactating women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2023-12-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
ORR | up to 2 years
  Objective response rate by INV assessment per RECIST
PFS | from the first dose until firstly confirmed and recorded disease progression or death (whichever occurs earlier),assessed up to 2 years
  Progression-free survival by INV assessment per RECIST

SECONDARY OUTCOMES:
OS | from the date of first dose unitl the date of death from any cause, assessed up to 2 years
  Overall survival
DOR | from the date when CR or PR (whichever recorded earlier) is firstly achieved until the date when disease progression or death is firstly recorded (whichever occurs earlier),assessed up to 2 years
  Duration of response